CLINICAL TRIAL: NCT06546774
Title: The Effect of Melatonin Supplementation on Cumulus Cells and Reproductive Outcomes in Older Women Undergoing IVF Cycles
Brief Title: The Effect of Melatonin Supplementation on Cumulus Cells and IVF Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Li-Te Lin, Attending doctor, Department of Obstetrics and Gynecology, Principal Investigator, Associate professor, Kaohsiung Veterans General Hospital.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSVGH21-CT1-43
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Unrecognized Condition
Keywords: Melatonin; Cumulus cells; In vitro fertilization; Old women; Infertility
MeSH Terms: conditions — Infertility | interventions — Melatonin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin group (Experimental): Patients received melatonin supplementation for at least a two-month period prior to IVF cycles
  Interventions: Dietary Supplement: Melatonin
- Control group (No Intervention): Patients did not receive melatonin supplementation and proceeded directly to IVF cycles

INTERVENTIONS:
Dietary Supplement: Melatonin — In the study group, patients will receive melatonin supplementation for at least two months prior to IVF cycles
  Arms: Melatonin group

SUMMARY:
This study investigates the effects of melatonin supplementation on cumulus cell gene expression and in vitro fertilization (IVF) outcomes in women over 35 years old. In the study group, patients will receive melatonin supplementation for at least two months prior to their IVF cycles. Cumulus cells will be collected after oocyte retrieval, and IVF outcomes will be assessed.

DETAILED DESCRIPTION:
Aging in female reproductive cells, particularly cumulus granulosa cells, is associated with various dysfunctions that compromise fertility. Melatonin, a hormone primarily produced by the pineal gland, is renowned for its multifaceted roles in regulating physiological processes, including sleep-wake cycles, immune function, and antioxidative defense. Melatonin's antioxidant action is mediated through direct scavenging of free radicals, upregulation of antioxidant enzymes, and improvement of mitochondrial efficiency. These properties make melatonin a promising candidate for mitigating the adverse effects of aging on cellular function. This study aims to explore the effects of melatonin supplementation on cumulus cell gene expression and in vitro fertilization (IVF) outcomes in women over 35 years old. In the study group, patients will receive melatonin supplementation for at least two months prior to their IVF cycles. In the control group, patients will proceed directly to IVF cycles without melatonin supplementation. Cumulus cells will be collected after oocyte retrieval, and gene expression will be measured. Additionally, clinical pregnancy rate, live birth rate, and miscarriage rate between the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-45 years
* BMI 18-30 kg/m2
* planning to undergo IVF cycles

Exclusion Criteria:

* Primary ovarian insufficiency
* history of oophorectomy
* receiving oocyte donation
* Chromosome anomaly
* Congenital uterine anomaly
* Severe intrauterine adhesion
* Malignancy
* Using hormone therapy or supplements in recent 3 months

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Infertile women planning to undergo IVF cycles
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate (%) | through study completion, an average of 4 year
  a viable infant after 24 weeks of gestation
oxygen consumption rate of mitochodria (%) | through study completion, an average of 4 year
  to assess mitocondrial function in cumulus cells
mRNA levels of cumulus cell genes | through study completion, an average of 4 year
  to assess cumulus cells gene expression analysis

SECONDARY OUTCOMES:
Clinical pregnancy rate (%) | through study completion, an average of 4 year
  the presence of a fetal heartbeat detected via transvaginal sonography at 6-7 weeks of gestation
Ongoing pregnancy rate (%) | through study completion, an average of 4 year
  the continuation of the pregnancy beyond 12 weeks of gestation
Amount of ATP production (moles/min) of mitochodria | through study completion, an average of 4 year
  to assess mitocondrial function in cumulus cells

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Hao Tsui, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Department of Obstetrics and Gynecology, Kaohsiung Veterans General Hospital, Kaohsiung, Taiwan, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kandil OM, Rahman SMAE, Ali RS, Ismail EA, Ibrahim NM. Effect of melatonin on developmental competence, mitochondrial distribution, and intensity of fresh and vitrified/thawed in vitro matured buffalo oocytes. Reprod Biol Endocrinol. 2024 Apr 5;22(1):39. doi: 10.1186/s12958-024-01209-7. PMID 38580962
- [Result] Navid S, Saadatian Z, Talebi A. Assessment of developmental rate of mouse embryos yielded from in vitro fertilization of the oocyte with treatment of melatonin and vitamin C simultaneously. BMC Womens Health. 2023 Oct 4;23(1):525. doi: 10.1186/s12905-023-02673-w. PMID 37794412
- [Result] He C, Wang J, Zhang Z, Yang M, Li Y, Tian X, Ma T, Tao J, Zhu K, Song Y, Ji P, Liu G. Mitochondria Synthesize Melatonin to Ameliorate Its Function and Improve Mice Oocyte's Quality under in Vitro Conditions. Int J Mol Sci. 2016 Jun 14;17(6):939. doi: 10.3390/ijms17060939. PMID 27314334
- [Result] Yang M, Tao J, Chai M, Wu H, Wang J, Li G, He C, Xie L, Ji P, Dai Y, Yang L, Liu G. Melatonin Improves the Quality of Inferior Bovine Oocytes and Promoted Their Subsequent IVF Embryo Development: Mechanisms and Results. Molecules. 2017 Nov 27;22(12):2059. doi: 10.3390/molecules22122059. PMID 29186876
- [Result] Zhao XM, Wang N, Hao HS, Li CY, Zhao YH, Yan CL, Wang HY, Du WH, Wang D, Liu Y, Pang YW, Zhu HB. Melatonin improves the fertilization capacity and developmental ability of bovine oocytes by regulating cytoplasmic maturation events. J Pineal Res. 2018 Jan;64(1). doi: 10.1111/jpi.12445. Epub 2017 Oct 11. PMID 28833478
- [Result] Dai X, Lu Y, Zhang M, Miao Y, Zhou C, Cui Z, Xiong B. Melatonin improves the fertilization ability of post-ovulatory aged mouse oocytes by stabilizing ovastacin and Juno to promote sperm binding and fusion. Hum Reprod. 2017 Mar 1;32(3):598-606. doi: 10.1093/humrep/dew362. PMID 28137755
- [Result] Miao Y, Zhou C, Bai Q, Cui Z, ShiYang X, Lu Y, Zhang M, Dai X, Xiong B. The protective role of melatonin in porcine oocyte meiotic failure caused by the exposure to benzo(a)pyrene. Hum Reprod. 2018 Jan 1;33(1):116-127. doi: 10.1093/humrep/dex331. PMID 29112712
- [Result] Zhang M, Dai X, Lu Y, Miao Y, Zhou C, Cui Z, Liu H, Xiong B. Melatonin protects oocyte quality from Bisphenol A-induced deterioration in the mouse. J Pineal Res. 2017 Apr;62(3). doi: 10.1111/jpi.12396. Epub 2017 Mar 1. PMID 28178360
- [Result] Wei D, Zhang C, Xie J, Song X, Yin B, Liu Q, Hu L, Hao H, Geng J, Wang P. Supplementation with low concentrations of melatonin improves nuclear maturation of human oocytes in vitro. J Assist Reprod Genet. 2013 Jul;30(7):933-8. doi: 10.1007/s10815-013-0021-2. Epub 2013 Jun 6. PMID 23737216
- [Result] Bao Z, Li G, Wang R, Xue S, Zeng Y, Deng S. Melatonin Improves Quality of Repeated-Poor and Frozen-Thawed Embryos in Human, a Prospective Clinical Trial. Front Endocrinol (Lausanne). 2022 May 13;13:853999. doi: 10.3389/fendo.2022.853999. eCollection 2022. PMID 35634513
- [Result] Nishihara T, Hashimoto S, Ito K, Nakaoka Y, Matsumoto K, Hosoi Y, Morimoto Y. Oral melatonin supplementation improves oocyte and embryo quality in women undergoing in vitro fertilization-embryo transfer. Gynecol Endocrinol. 2014 May;30(5):359-62. doi: 10.3109/09513590.2013.879856. Epub 2014 Mar 17. PMID 24628045
- [Result] Eryilmaz OG, Devran A, Sarikaya E, Aksakal FN, Mollamahmutoglu L, Cicek N. Melatonin improves the oocyte and the embryo in IVF patients with sleep disturbances, but does not improve the sleeping problems. J Assist Reprod Genet. 2011 Sep;28(9):815-20. doi: 10.1007/s10815-011-9604-y. Epub 2011 Jul 12. PMID 21748445
- [Result] Batioglu AS, Sahin U, Gurlek B, Ozturk N, Unsal E. The efficacy of melatonin administration on oocyte quality. Gynecol Endocrinol. 2012 Feb;28(2):91-3. doi: 10.3109/09513590.2011.589925. Epub 2011 Jul 20. PMID 21770829
- [Result] Jahromi BN, Sadeghi S, Alipour S, Parsanezhad ME, Alamdarloo SM. Effect of Melatonin on the Outcome of Assisted Reproductive Technique Cycles in Women with Diminished Ovarian Reserve: A Double-Blinded Randomized Clinical Trial. Iran J Med Sci. 2017 Jan;42(1):73-78. PMID 28293053
- [Result] Hu KL, Ye X, Wang S, Zhang D. Melatonin Application in Assisted Reproductive Technology: A Systematic Review and Meta-Analysis of Randomized Trials. Front Endocrinol (Lausanne). 2020 Mar 27;11:160. doi: 10.3389/fendo.2020.00160. eCollection 2020. PMID 32292388
- [Result] Mejlhede MAB, Jepsen JB, Knudsen UB. Oral melatonin supplementation during in vitro fertilization treatment: a systematic PRISMA review and meta-analysis of randomized controlled trials. Gynecol Endocrinol. 2021 Dec;37(12):1079-1085. doi: 10.1080/09513590.2021.1974378. Epub 2021 Sep 8. PMID 34494508